CLINICAL TRIAL: NCT04813770
Title: The Impact of Theory-based Messaging on Covid-19 Vaccination Intentions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Katie Robb, Reader, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 200200052
Record Dates: First submitted 2021-03-23; First posted 2021-03-24 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Vaccination; Covid19
Keywords: vaccine hesitancy; vaccination uptake; messaging; illness beliefs; treatment beliefs
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Participants will not be blinded to the assigned intervention but will not be informed of the purpose of the study until they have completed the follow-up survey, at which point they will be debriefed. Investigators will be blinded to allocation because all procedures will be undertaken digitally and remotely without any investigator contact with participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theory-based messages (Experimental): Theory-based health messages about COVID-19 and COVID-19 vaccination, the necessity of COVID-19 vaccination to oneself and others, and COVID-19 vaccine regulatory approval processes. These messages are based on publicly available information and are hypothesised to increase perceived necessity and reduce concerns about vaccination, and target known barriers to vaccine uptake.
  Interventions: Behavioral: Theory-based messages
- General messages (Active Comparator): General messages about the COVID-19 virus and the vaccination programme. These messages do not target necessity and concerns, but are anticipated to promote understanding of the pandemic.
  Interventions: Behavioral: General messages

INTERVENTIONS:
Behavioral: Theory-based messages — COVID-19 vaccination information structured to address vaccination necessity and concerns.
  Arms: Theory-based messages
Behavioral: General messages — General messages about the COVID-19 virus and the vaccination programme.
  Arms: General messages

SUMMARY:
Uptake of vaccination against COVID-19 is key to controlling the pandemic. However, a significant proportion of people report that they do not intend to have a vaccine, often because of concerns they have about its side effects or safety. It is important to identify ways to communicate information about the vaccines that facilitate informed decisions rather than promoting uptake through coercion. This study will assess whether theory-based messages can change beliefs and increase intentions to receive a COVID-19 vaccine in Scotland. The messages will be based on publicly available information about the need for COVID-19 vaccination and the safety of the vaccines, and structured to address specific types of treatment beliefs. Participants will be randomised to either a group shown the messages or a control group shown general information messages about the COVID-19 virus and vaccination programme. By comparing the two groups we aim to test what impact the theory-based messages have on intentions and beliefs about COVID-19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial
* Aged 18 years or above
* Resident in Scotland

Exclusion Criteria:

* Received at least one COVID-19 vaccination dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1113 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Covid-19 vaccination intention measured by a single item and aggregated as the proportion of intenders. | Immediately post-intervention
  Participants will be asked: "If you were invited to have a COVID-19 vaccination would you take the vaccine?" Those responding "yes, probably" or "yes, definitely" will be treated as intenders. Those responding "don't know", "probably not" or "definitely not" will be treated as non-intenders.

SECONDARY OUTCOMES:
Mean COVID-19 illness coherence score as assessed by the IPQ-R | Immediately post-intervention
  Self-reported COVID-19 illness coherence as assessed by the the illness coherence subscale of the revised Illness Perception Questionnaire (IPQ-R), with a minimum score of 5, a maximum score of 25 and a higher score representing greater personal understanding of COVID-19.
Mean perceived necessity score as assessed by the BMQ | Immediately post-intervention
  Self-reported perceived necessity of a COVID-19 vaccine as assessed by the Specific-Necessity subscale of the Beliefs about Medicines Questionnaire (BMQ), with a minimum score of 5, a maximum score of 25 and a higher score representing greater perceived necessity of a COVID-19 vaccine.
Mean perceived concerns score as assessed by the BMQ | Immediately post-intervention
  Self-reported perceived concerns about a COVID-19 vaccine as assessed by the Specific-Concerns subscale of the Beliefs about Medicines Questionnaire (BMQ), with a minimum score of 5, a maximum score of 25 and a higher score representing greater perceived concerns about a COVID-19 vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Robb, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual level study data will be shared via the University of Glasgow's repository Enlighten: Research Data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: On publication of the study results for a period of ten years.
Access Criteria: Data will be made publicly available.

REFERENCES:
- [Derived] Young B, Kotzur M, Gatting L, Bonner C, Ayre J, McConnachie A, Batcup C, McCaffery K, O'Carroll R, Robb KA. The impact of theory-based messages on COVID-19 vaccination intentions: a structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Apr 29;22(1):311. doi: 10.1186/s13063-021-05277-7. PMID 33926540